CLINICAL TRIAL: NCT00004918
Title: A Phase I/II Study of PR1 (NSC 698102) Human Leukemia Peptide Vaccine With Montanide ISA 51 (NSC 675756) or Montanide ISA 51 VG (NSC 737063) Adjuvant
Brief Title: Vaccine Therapy Plus Immune Adjuvant in Treating Patients With Chronic Myeloid Leukemia, Acute Myeloid Leukemia, or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03086; DM 97-325
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia in Remission; Chronic Phase Chronic Myelogenous Leukemia; Previously Treated Myelodysplastic Syndromes; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts | interventions — montanide ISA 51; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (3):
- Arm I (dose level 1 PR1 leukemia peptide vaccine) (Experimental): Patients receive dose level 1 of PR1 leukemia peptide vaccine with Montanide ISA-51 SC once every 3 weeks for 18 weeks, for a total of 6 vaccinations. Patients also receive GM-CSF SC with each vaccination.
  Interventions: Biological: PR1 leukemia peptide vaccine; Drug: Montanide ISA 51 VG; Biological: sargramostim; Other: laboratory biomarker analysis
- Arm II (dose level 2 PR1 leukemia peptide vaccine) (Experimental): Patients receive dose level 2 of PR1 leukemia peptide vaccine with Montanide ISA-51 SC once every 3 weeks for 18 weeks, for a total of 6 vaccinations. Patients also receive GM-CSF SC with each vaccination.
  Interventions: Biological: PR1 leukemia peptide vaccine; Drug: Montanide ISA 51 VG; Biological: sargramostim; Other: laboratory biomarker analysis
- Arm III (dose level 3 PR1 leukemia peptide vaccine) (Experimental): Patients receive dose level 3 of PR1 leukemia peptide vaccine with Montanide ISA-51 SC once every 3 weeks for 18 weeks, for a total of 6 vaccinations. Patients also receive GM-CSF SC with each vaccination.
  Interventions: Biological: PR1 leukemia peptide vaccine; Drug: Montanide ISA 51 VG; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: PR1 leukemia peptide vaccine — Given SC
  Other Names: PR1 vac; proteinase 3 PR1 peptide
Drug: Montanide ISA 51 VG — Given SC
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Vaccines made from peptides that are found on leukemia cells may make the body build an immune response and kill cancer cells. Combining vaccine therapy with the immune adjuvant Montanide ISA-51 may be a more effective treatment for chronic myeloid leukemia, acute myeloid leukemia, or myelodysplastic syndrome. This phase I/II trial is studying the side effects and best dose of vaccine therapy when given with Montanide ISA-51 and to see how well they work in treating patients with chronic myeloid leukemia, acute myeloid leukemia, or myelodysplastic syndrome

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate both toxicity and immune response efficacy of PR1 peptide (PR1 leukemia peptide vaccine) administered subcutaneously.

SECONDARY OBJECTIVES:

I. To evaluate possible clinical efficacy of PR1 peptide vaccine preparation with Montanide ISA 51 or Montanide ISA 51 VG adjuvant, in high-risk HLA-A2 positive patients with myeloid leukemias.

OUTLINE: This is a phase I dose-escalation study of PR1 leukemia peptide vaccine, followed by a phase II randomized study.

Patients receive PR1 leukemia peptide vaccine with Montanide ISA-51 (ISA-51) subcutaneously (SC) once every 3 weeks for 18 weeks, for a total of 6 vaccinations. Patients also receive sargramostim (GM-CSF) SC with each vaccination.

Cohorts of 3 patients receive escalating doses of PR1 leukemia peptide vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity.

Additional patients are accrued to the phase II portion of the study and are randomized to receive one of three dose levels of PR1 leukemia peptide vaccine with ISA-51. Patients in each of the 3 arms receive treatment as in the phase I portion of the study.

Patients achieving a clinical response and/or clinical response to the vaccine whose disease progresses within 6-12 months after the first set of vaccinations may receive additional vaccine as before.

Patients achieving a clinical response or immune reaction to the vaccine are followed at least monthly until death or until the clinical response and/or immune reaction is lost.

PROJECTED ACCRUAL: A total of 3-9 patients will be accrued for the phase I dose escalation portion of this study. A maximum of 60 patients (20 per arm) will be accrued for the phase II randomized portion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be HLA-A2 positive at one allele
* Patients with CML in chronic phase or early accelerated phase, who are not eligible for BMT or interferon, or have failed standard therapy, or have relapsed after BMT
* Patients with MDS (FAB subtypes RAEB, and RAEBt) or AML in second or subsequent remission, or AML with a smoldering presentation and who are not candidates for chemotherapy, and who are believed to have a life expectancy of at least 9 weeks
* ECOG performance status < 3
* Life expectancy is not severely limited by concomitant illness
* Serum bilirubin < 3 mg/dl
* Serum creatinine < 2 mg/dl
* ALT < 3 x the upper limit of normal
* No serologic antibody against proteinase 3
* No known history of Wegener's granulomatosis or other vasculitis
* FEV, FVC, and DLCO > 50% of predicted, and no symptomatic pulmonary disease
* Not pregnant; all female patients will have a serum pregnancy test, and only those that test negative will be allowed on study
* HIV negative
* No known allergic reaction to Montanide ISA 51 or Montanide ISA 51 VG adjuvant
* No active uncontrolled infection
* Patient or representative able to understand the study and consent
* Patient is not receiving steroids, cyclosporine, or FK-506 for at least 1 month prior to study entry and during study period
* No concomitant use of interferon or chemotherapy during study period other than hydroxyurea to control cell counts
* Patients who relapsed within one year of completing the initial vaccination could be retreated with up to 6 additional vaccinations if they remain eligible for treatment according to the original criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 1999-12; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adverse event DTOX (death or autoimmune toxicity or vascular toxicity at any time) assessed using Common Toxicity Criteria (CTC) version 2.0 | Up to 8 years
Ability of dose | Up to 8 years
  Regression analyses will be performed.
T cell receptor (TCR) activity | Up to 8 years
  Regression analyses will be performed.
Clinical response | Up to 8 years
  Regression analyses will be performed.
Duration of first immune response (IR) | Up to 8 years
  Will be assessed using logistic regression.
Survival time | Up to 8 years
  Will be assessed using a Cox model or similar event time model

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar Qazilbash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States